CLINICAL TRIAL: NCT03743402
Title: Randomized Trial of Telephonic Pain Self-management to Promote Opioid Tapering
Brief Title: Strategies to Improve Pain and Enjoy Life
Acronym: STRIPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Kaiser Permanente (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Mark Sullivan, Professor of Psychiatry and Behavioral Sciences, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SITE00000193; R01DA044970-01 (NIH)
Record Dates: First submitted 2018-10-09; First posted 2018-11-16 (Actual); Results first posted 2023-04-07 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Chronic Pain
Keywords: long-term opioid therapy; chronic pain self-management; primary care prescribing guidance
MeSH Terms: conditions — Chronic Pain | interventions — Motivational Interviewing; Physicians, Primary Care

STUDY DESIGN:
Intervention Model Description: Patients are individually randomized to pain self-management training for opioid taper or usual care. Those randomized to pain self-management training will be offered assistance with opioid taper during approximately the fourth session of pain self-management training.
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessment will be conducted by Kaiser survey team which will be blind to treatment assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pain self-management (Experimental): This intervention will have 4 components:
  1. telephone-delivered evidence-based pain self-management training,
  2. web-based video of successfully tapered patients with motivational interviewing debriefing,
  3. a voluntary, self-paced opioid taper
  4. opioid and non-opioid prescribing guidance for the patient's primary care provider.
  Interventions: Behavioral: Pain self-management training; Behavioral: video education, motivational interviewing; Behavioral: voluntary self-paced opioid taper; Behavioral: prescribing guidance for primary care provider
- usual care (Active Comparator): Patients randomized to usual care will continue to receive care as usual from their Kaiser primary care provider.
  Interventions: Other: usual care

INTERVENTIONS:
Behavioral: Pain self-management training — This intervention will have 4 components:
  1. telephone-delivered evidence-based pain self-management training,
  2. web-based video of successfully tapered patients with motivational interviewing debriefing,
  3. a voluntary, self-paced opioid taper
  4. opioid and non-opioid prescribing guidance for the patient's primary care provider.
  Other Names: phone cognitive-behavioral pain self-management training
  Arms: Pain self-management
Behavioral: video education, motivational interviewing — web-based video of successfully tapered patients with motivational interviewing debriefing
  Other Names: exposure to successfully tapered patients with debriefing
  Arms: Pain self-management
Behavioral: voluntary self-paced opioid taper — Voluntary self-paced opioid taper where patient chooses whether, when and how much to taper opioids. Taper schedule and strategy will be proposed to patients, but they will negotiate details with their primary care provider.
  Other Names: opioid daily dose reduction
  Arms: Pain self-management
Behavioral: prescribing guidance for primary care provider — Based upon review of medications and diagnoses in the electronic medical record, the principal investigator will offer guidance on opioid taper rate and strategy. He will also offer suggestions to adjust or initiate other psychotropic medications to treat pain or psychiatric comorbid illness that may be unmasked through opioid taper. All prescriptions will be written by the primary care provider.
  Other Names: medication initiation and adjustment suggestions to optimize control of pain and psychiatric comorbidity
  Arms: Pain self-management
Other: usual care — Usual care will consist of any and all regular care that may be offered by primary care for chronic pain and related illnesses
  Other Names: standard opioid therapy for chronic pain
  Arms: usual care

SUMMARY:
In the Strategies to Improve Pain and Enjoy Life (STRIPE) study, the effectiveness of a multicomponent intervention will be tested, compared with usual care, on opioid dose and pain outcomes among patients on high dose (≥ 40 mg morphine equivalent dose) long-term opioid therapy in a randomized controlled trial. This intervention will have 4 components: a) telephone-delivered evidence-based pain self-management training, b) web-based video of successfully tapered patients with motivational interviewing debriefing, c) a voluntary, self-paced opioid taper, and d) opioid and non-opioid prescribing guidance for the patient's primary care provider.

DETAILED DESCRIPTION:
In a National Institute on Drug Abuse-funded R34 pilot study of pain self-management training for prescription opioid taper support, it was demonstrated that 22 weeks of opioid taper support promotes opioid dose reduction more effectively than usual care (43% vs 19% dose reduction from baseline) with no increase in pain intensity and significantly reduced activity interference. This intervention will now be adapted and tested in a large integrated primary care system. To address patients' fears of opioid taper that limited recruitment into this pilot study, subjects will be randomized to pain self-management training and then offered the option of self-paced opioid taper. Specifically, the effectiveness of this intervention will be tested, compared with usual care, on opioid dose and pain outcomes among patients on moderate-high dose (≥ 40mg morphine equivalent dose) long-term opioid therapy (LtOT) in a randomized controlled trial. This intervention will have 4 components: a) telephone-delivered evidence-based pain self-management training, b) web-based video of successfully tapered patients with motivational interviewing debriefing, c) a voluntary, self-paced opioid taper, and d) opioid and non-opioid prescribing guidance for the patient's primary care provider. Specific Aim 1: To adapt a previously developed prescription opioid taper support intervention into a telephone-delivered pain self-management training that provides the option for supported opioid taper. This will be delivered in multiple primary care clinics by a nurse interventionist trained and supervised by a pain psychologist and will include guidance in opioid and non-opioid medication prescribing. Specific Aim 2: To test in a randomized trial the effects of this intervention on: a) opioid outcomes: daily opioid dose (primary outcome), percent dose reduction from baseline, problem opioid use (questionnaire and electronic health record text indicators), and patient-reported opioid difficulties; and b) pain-related outcomes: PEG (self-report of Pain intensity, Enjoyment of life interference, General activity interference; primary outcome), pain self-efficacy, and anxiety and depression symptoms. Hypotheses pertaining to opioid use: Patients receiving LtOT for chronic non-cancer pain (CNCP) randomized to the STRIPE intervention, as compared with those randomized to usual care, will have lower opioid doses, greater percent reduction of opioid dose, lower proportions with problem opioid use, lower opioid craving, and lower levels of patient-reported opioid-related difficulties at 6 and 12 months after randomization. Hypotheses pertaining to pain outcomes: Patients receiving LtOT for CNCP randomized to the STRIPE intervention, as compared with those randomized to usual care, will have lower PEG scores, higher levels of pain self-efficacy, higher global impression of change, and lower levels of anxiety and depressive symptoms at 6 and 12 months after randomization. The proposed trial will determine whether pain self-management training can promote prescription opioid taper in moderate-higher-dose long-term opioid therapy patients without increasing pain level or activity and enjoyment interference. If this trial is successful, then prescribers and patients may be able to pursue supported opioid taper without fear of escalating pain.

ELIGIBILITY:
Inclusion Criteria:

* age 18-80 years
* receiving care at a Kaiser Washington primary care clinic;
* Chronic Non-Cancer Pain, defined as patient-reported pain on more than half the days in the past 6 months;
* currently on higher-dose long-term opioid therapy, defined as >90 days' supply in the past 180 days with a mean daily dose of 40 mg MED or greater in the past 90 days, as first identified via Kaiser's pharmacy dispensing data and subsequently validated by patient self-report during screening for the trial
* consent to participate in the study arm to which they are randomly assigned
* able to read, speak, and write English adequate for outcome measures
* enrollment in Kaiser for at least 6 months prior and no plans to disenroll over the next year.

Exclusion Criteria:

* receiving treatment for cancer
* enrollment in palliative or hospice care
* use in past year of parenteral, transdermal, or transmucosal opioids
* residing in nursing home or assisted living
* using any implanted device for pain control
* psychotic symptoms, psychiatric hospitalization or suicide attempts in the past year
* current suicidal ideation with plan or intent
* dementia diagnosis in Electronic Health Record
* Patients on buprenorphine for any reason, or methadone or naltrexone for treatment of Opioid Use Disorder

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2019-04-04 (Actual); Primary Completion 2022-01-27 (Actual); Study Completion 2022-01-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark D Sullivan, MD, PhD, Principal Investigator — University of Washington
Locations (1):
- Kaiser Permanente Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
Availability of data and materials: The datasets generated and analyzed during the current study are not publicly available to protect participant privacy. Deidentified analysis datasets may be made available upon email request to the corresponding author. Any data shared may require an application with description of the planned research purpose and an execution of a data use agreement with approval from the KPWA IRB overseeing this trial. Further, if the researcher would also like the R analysis code used for this manuscript, they can request this at the time of requesting the deidentified analysis dataset.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available after January 30, 2023 until January 30, 2028
Access Criteria: Availability of data and materials: The datasets generated and analyzed during the current study are not publicly available to protect participant privacy. Deidentified analysis datasets may be made available upon email request to the corresponding author. Any data shared may require an application with description of the planned research purpose and an execution of a data use agreement with approval from the KPWA IRB overseeing this trial. Further, if the researcher would also like the R analysis code used for this manuscript, they can request this at the time of requesting the deidentified analysis dataset.

REFERENCES:
- [Background] Sullivan MD, Turner JA, DiLodovico C, D'Appollonio A, Stephens K, Chan YF. Prescription Opioid Taper Support for Outpatients With Chronic Pain: A Randomized Controlled Trial. J Pain. 2017 Mar;18(3):308-318. doi: 10.1016/j.jpain.2016.11.003. Epub 2016 Nov 28. PMID 27908840
- [Derived] Wartko PD, Krakauer C, Turner JA, Cook AJ, Boudreau DM, Sullivan MD. STRategies to Improve Pain and Enjoy life (STRIPE): results of a pragmatic randomized trial of pain coping skills training and opioid medication taper guidance for patients on long-term opioid therapy. Pain. 2023 Dec 1;164(12):2852-2864. doi: 10.1097/j.pain.0000000000002982. Epub 2023 Aug 25. PMID 37624901
- [Derived] Wartko PD, Boudreau DM, Turner JA, Cook AJ, Wellman RD, Fujii MM, Garcia RC, Moser KA, Sullivan MD. STRategies to Improve Pain and Enjoy life (STRIPE): Protocol for a pragmatic randomized trial of pain coping skills training and opioid medication taper guidance for patients on long-term opioid therapy. Contemp Clin Trials. 2021 Nov;110:106499. doi: 10.1016/j.cct.2021.106499. Epub 2021 Jul 2. PMID 34217889

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Using electronic health records and claims data, 1381 individuals fulfilled a subset of study inclusion criteria and were contacted to assess further inclusion criteria. 170 of these individuals fulfilled all inclusion criteria, as determined using two phone screenings and were contacted to participate in the study. 153 of these individuals returned a baseline questionnaire and were randomized.
Groups:
- Pain Self-Management: This arm includes patients randomized to Pain Self-Management Training. This intervention has 4 components:
  1. telephone-delivered evidence-based pain self-management training,
  2. web-based video of successfully tapered patients with motivational interviewing debriefing,
  3. a voluntary, self-paced opioid taper, and
  4. opioid and non-opioid prescribing guidance for the patient's primary care provider.
Period: Overall Study
Arm/Group | Pain Self-Management | Usual Care
Started | 79 | 74
Availability of at Least One Primary Outcome Measure at 6 Months Post-baseline | 79 | 74
Completed (Defined to be availability of at least one primary outcome measure at 12 months post-baseline.) | 78 | 73
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pain Self-Management | Usual Care | Total
Number analyzed (Participants) | 79 | 74 | 153
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.7 (10.7) | 60.7 (10.6) | 60.7 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 45 | 98
  Male | 26 | 29 | 55
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 3
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 2
  Black or African American | 1 | 6 | 7
  White | 64 | 62 | 126
  More than one race | 3 | 2 | 5
  Unknown or Not Reported | 6 | 3 | 9
Region of Enrollment [Number; unit: participants]
  United States | 79 | 74 | 153
Daily Opioid Morphine Milligram Equivalents (MME) [Mean (Standard Deviation); unit: MME/day] — Average over the 30 days prior to baseline of the prescribed daily morphine milligram equivalents (MME).
  MME/day | 77.1 (67.9) | 72.8 (30.3) | 75.0 (53.0)
Pain, Enjoyment of Life, and General Activity (PEG) Score [Mean (Standard Deviation); unit: score on a scale] — A 3-item, self-report measure reflecting average pain intensity, pain interference with general activity, and pain interference with enjoyment of life in the past week. It is scored on a scale of 0 to 10; higher scores indicate worse pain intensity and interference with life and enjoyment of activities.
  score on a scale | 6.5 (1.8) | 6.6 (1.8) | 6.6 (1.8)
Pain Self-Efficacy Questionnaire (PSEQ) Score [Mean (Standard Deviation); unit: score on a scale] — Score from a 10-item questionnaire about pain self-efficacy that range between 0 and 60; higher scores indicate higher confidence in ability to do activities despite pain.
  score on a scale | 29.9 (10.4) | 27.7 (13.0) | 28.8 (11.8)
Patient Health Questionnaire-8 (PHQ-8) Score [Mean (Standard Deviation); unit: score on a scale] — An 8-item questionnaire used to assess depression with scores between 0 and 24; higher scores indicate greater depression severity.
  score on a scale | 8.1 (5.1) | 8.8 (4.7) | 8.5 (4.9)
Generalized Anxiety Disorder-7 (GAD-7) Score [Mean (Standard Deviation); unit: score on a scale] — A 7-item questionnaire used to assess anxiety with scores between 0 and 21; higher scores indicate greater anxiety severity.
  score on a scale | 4.7 (4.8) | 5.3 (4.5) | 5.0 (4.6)
Prescription Opioid Misuse Index (POMI) Score [Mean (Standard Deviation); unit: score on a scale] — A 6-item questionnaire used to assess problem opioid use with scores between 0 and 6; higher scores indicate a greater likelihood of having opioid use disorder.
  score on a scale | 0.7 (0.9) | 0.8 (0.9) | 0.7 (0.9)
Prescribed Opioids Difficulties Scale (PODS) Score [Mean (Standard Deviation); unit: score on a scale] — A 15-item questionnaire used to assess patient-perceived difficulties and concerns attributed to the use of opioid medication with scores between 0 and 60; higher scores indicate greater difficulties and concerns.
  score on a scale | 9.3 (7.5) | 10.5 (8.1) | 9.9 (7.8)
Opioid Craving Score [Mean (Standard Deviation); unit: score on a scale] — A single-item questionnaire used to assess opioid craving in the past week with scores between 0 and 10; higher scores indicate greater craving.
  score on a scale | 1.0 (2.1) | 1.5 (2.8) | 1.3 (2.5)

OUTCOME MEASURES:

1. Primary Outcome: Daily Opioid Morphine Milligram Equivalents (MME)
Description: Average over the prior 30 days of the prescribed daily morphine milligram equivalents (MME).
Time Frame: 12 months after randomization
Population: Randomized individuals with complete electronic prescription records available during the 6- and/or 12-month post-randomization assessment period with non-missing baseline data used for adjustment in regression models.
Measure: Mean (95% Confidence Interval); unit: MME/day
Arm/Group | Pain Self-Management | Usual Care
Number analyzed (Participants) | 75 | 72
MME/day | 65.17 [58.86 to 71.49] | 67.51 [62.49 to 72.54]
Statistical Analysis 1: Comparison: Pain Self-Management vs Usual Care; A priori power calculations indicated 90% power to detect an average 24 MME/day difference between arms; Test type: Equivalence — The null hypothesis was a point null of exactly 0 expected difference in MME/day between arms; p = 0.58, Regression, Linear; Mean Difference (Final Values) = -2.54, 95% CI 2-sided [-10.55 to 5.88] — mean difference=(pain self-management)-(usual care)

2. Primary Outcome: Pain, Enjoyment of Life, and General Activity (PEG) Score
Description: A 3-item, self-report measure reflecting average pain intensity, pain interference with general activity, and pain interference with enjoyment of life in the past week. It is scored on a scale of 0 to 10; higher scores indicate worse pain intensity and interference with life and enjoyment of activities.
Time Frame: 12 months after randomization
Population: Randomized individuals who completed the 6-month and/or 12-month PEG questionnaire and with complete baseline data used for adjustment in regression models.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Pain Self-Management | Usual Care
Number analyzed (Participants) | 64 | 71
score on a scale | 6.14 [5.79 to 6.49] | 6.14 [5.76 to 6.51]
Statistical Analysis 1: Comparison: Pain Self-Management vs Usual Care; A priori power calculations indicated 90% power to detect a 1.2-point average difference in PEG score between arms; Test type: Equivalence — The null hypothesis was a point null of exactly 0 expected difference in PEG score between arms; p = 0.98, Regression, Linear; Mean Difference (Final Values) = 0.01, 95% CI 2-sided [-0.51 to 0.52] — mean difference = (pain self-management)-(usual care)

3. Secondary Outcome: Daily Opioid Morphine Milligram Equivalents (MME)
Description: Average over the prior 30 days of the prescribed daily morphine milligram equivalents (MME).
Time Frame: 6 months after randomization
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: MME/day
Arm/Group | Pain Self-Management | Usual Care
Number analyzed (Participants) | 75 | 72
MME/day | 73.03 [67.65 to 78.42] | 71.74 [67.37 to 76.11]
Statistical Analysis 1: Comparison: Pain Self-Management vs Usual Care; Test type: Equivalence — The null hypothesis was a point null of exactly 0 difference in average MME/day between arms; p = 0.72, Regression, Linear; Mean Difference (Final Values) = 1.30, 95% CI 2-sided [-5.69 to 8.29] — mean difference=(pain self-management)-(usual care)

4. Secondary Outcome: Pain, Enjoyment of Life, and General Activity (PEG) Score
Description: as for outcome 2
Time Frame: 6 months after randomization
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Pain Self-Management | Usual Care
Number analyzed (Participants) | 64 | 71
score on a scale | 6.06 [5.63 to 6.49] | 6.59 [6.22 to 6.95]
Statistical Analysis 1: Comparison: Pain Self-Management vs Usual Care; Test type: Equivalence — The null hypothesis is a point null of exactly 0 difference in expected PEG score between arms; p = 0.07, Regression, Linear; Mean Difference (Final Values) = -0.53, 95% CI 2-sided [-1.11 to 0.05] — mean difference = (pain self-management) - (usual care)

5. Secondary Outcome: Pain Self-Efficacy Questionnaire (PSEQ) Score
Description: Score from a 10-item questionnaire about pain self-efficacy that range between 0 and 60; higher scores indicate higher confidence in ability to do activities despite pain.
Time Frame: 6 months after randomization
Population: Randomized individuals with completed PSEQ questionnaires at 6- and/or 12-months post-randomization with non-missing baseline data used for adjustment in regression models.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Pain Self-Management | Usual Care
Number analyzed (Participants) | 62 | 69
score on a scale | 32.31 [8.61 to 56.01] | 30.21 [22.06 to 38.35]
Statistical Analysis 1: Comparison: Pain Self-Management vs Usual Care; Test type: Equivalence — The null hypothesis is a point null of exactly 0 expected difference in PSEQ score between arms; p = 0.80, Regression, Linear; Mean Difference (Final Values) = 2.11, 95% CI 2-sided [-13.83 to 18.04] — mean difference = (pain self-management) - (usual care)

6. Secondary Outcome: Pain Self-Efficacy Questionnaire (PSEQ) Score
Description: as for outcome 5
Time Frame: 12 months after randomization
Population: as for outcome 5
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Pain Self-Management | Usual Care
Number analyzed (Participants) | 62 | 69
score on a scale | 31.97 [19.47 to 44.47] | 27.65 [15.56 to 39.74]
Statistical Analysis 1: Comparison: Pain Self-Management vs Usual Care; Test type: Equivalence — The null hypothesis is a point null of exactly 0 expected difference in PSEQ score between arms; p = 0.02, Regression, Linear; Mean Difference (Final Values) = 4.33, 95% CI 2-sided [0.56 to 8.09] — mean difference = (pain self-management) - (usual care)

7. Secondary Outcome: Patient Health Questionnaire-8 (PHQ-8) Score
Description: An 8-item questionnaire used to assess depression with scores between 0 and 24; higher scores indicate greater depression severity.
Time Frame: 6 months after randomization
Population: Randomized individuals with completed PHQ-8 questionnaires at 6- and/or 12-months post-randomization with non-missing baseline data used for adjustment in regression models.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Pain Self-Management | Usual Care
Number analyzed (Participants) | 61 | 68
score on a scale | 8.25 [5.24 to 11.26] | 8.60 [7.19 to 10.01]
Statistical Analysis 1: Comparison: Pain Self-Management vs Usual Care; Test type: Equivalence — The null hypothesis is a point null of exactly 0 expected difference in PHQ-8 score between arms; p = 0.75, Regression, Linear; Mean Difference (Final Values) = -0.35, 95% CI 2-sided [-2.53 to 1.82] — mean difference = (pain self-management) - (usual care)

8. Secondary Outcome: Patient Health Questionnaire-8 (PHQ-8) Score
Description: as for outcome 7
Time Frame: 12 months after randomization
Population: as for outcome 5
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Pain Self-Management | Usual Care
Number analyzed (Participants) | 61 | 68
score on a scale | 7.54 [5.89 to 9.19] | 8.04 [6.33 to 9.75]
Statistical Analysis 1: Comparison: Pain Self-Management vs Usual Care; Test type: Equivalence — The null hypothesis is a point null of exactly 0 expected difference in PHQ-8 score between arms; p = 0.48, Regression, Linear; Mean Difference (Final Values) = -0.50, 95% CI 2-sided [-1.87 to 0.87] — mean difference = (pain self-management) - (usual care)

9. Secondary Outcome: Generalized Anxiety Disorders-7 (GAD-7) Score
Description: A 7-item questionnaire used to assess anxiety with scores between 0 and 21; higher scores indicate greater anxiety severity.
Time Frame: 6 months after randomization
Population: Randomized individuals with completed GAD-7 questionnaires at 6- and/or 12-months post-randomization with non-missing baseline data used for adjustment in regression models.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Pain Self-Management | Usual Care
Number analyzed (Participants) | 64 | 71
score on a scale | 4.89 [2.79 to 7.00] | 5.14 [3.57 to 6.72]
Statistical Analysis 1: Comparison: Pain Self-Management vs Usual Care; Test type: Equivalence — The null hypothesis is a point null of exactly 0 expected difference in GAD-7 score between arms; p = 0.64, Regression, Linear; Mean Difference (Final Values) = -0.25, 95% CI 2-sided [-1.31 to 0.81] — mean difference = (pain self-management) - (usual care)

10. Secondary Outcome: Generalized Anxiety Disorders-7 (GAD-7) Score
Description: as for outcome 9
Time Frame: 12 months after randomization
Population: as for outcome 9
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Pain Self-Management | Usual Care
Number analyzed (Participants) | 64 | 71
score on a scale | 5.20 [4.07 to 6.33] | 4.91 [4.03 to 5.80]
Statistical Analysis 1: Comparison: Pain Self-Management vs Usual Care; Test type: Equivalence — The null hypothesis is a point null of exactly 0 expected difference in GAD-7 score between arms; p = 0.65, Regression, Linear; Mean Difference (Final Values) = 0.28, 95% CI 2-sided [-0.94 to 1.51] — mean difference = (pain self-management) - (usual care)

11. Secondary Outcome: Patient Global Impression of Change (PGIC) Score
Description: Single 7-point scale assessing global improvement with treatment, range 0 (bad) - 7 (good)
Time Frame: 6 months after randomization
Population: Randomized individuals with completed PGIC questionnaires at 6- and/or 12-months post-randomization with non-missing baseline data used for adjustment in regression models.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Pain Self-Management | Usual Care
Number analyzed (Participants) | 64 | 71
score on a scale | 3.12 [2.76 to 3.47] | 2.51 [2.16 to 2.86]
Statistical Analysis 1: Comparison: Pain Self-Management vs Usual Care; Test type: Equivalence — The null hypothesis is a point null of exactly 0 expected difference in PGIC score between arms; p = 0.02, Regression, Linear; Mean Difference (Final Values) = 0.61, 95% CI 2-sided [0.12 to 1.10] — mean difference = (pain self-management) - (usual care)

12. Secondary Outcome: Patient Global Impression of Change (PGIC) Score
Description: Single 7-point scale assessing global improvement with treatment, range 0 (bad) - 7 (good)
Time Frame: 12 months after randomization
Population: as for outcome 11
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Pain Self-Management | Usual Care
Number analyzed (Participants) | 64 | 71
score on a scale | 3.71 [3.27 to 4.15] | 2.38 [2.04 to 2.73]
Statistical Analysis 1: Comparison: Pain Self-Management vs Usual Care; Test type: Equivalence — The null hypothesis is a point null of exactly 0 expected difference in PGIC score between arms; p < 0.01, Regression, Linear; Mean Difference (Final Values) = 1.33, 95% CI 2-sided [0.77 to 1.88] — mean difference = (pain self-management) - (usual care)

13. Secondary Outcome: Prescription Opioid Misuse Index (POMI) Score
Description: A 6-item questionnaire used to assess problem opioid use with scores between 0 and 6; higher scores indicate a greater likelihood of having opioid use disorder.
Time Frame: 6 months after randomization
Population: Randomized individuals with completed POMI questionnaires at 6- and/or 12-months post-randomization with non-missing baseline data used for adjustment in regression models.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Pain Self-Management | Usual Care
Number analyzed (Participants) | 64 | 69
score on a scale | 0.56 [0.38 to 0.74] | 0.47 [0.33 to 0.61]
Statistical Analysis 1: Comparison: Pain Self-Management vs Usual Care; Test type: Equivalence — The null hypothesis is a point null of exactly 0 expected difference in POMI score between arms; p = 0.42, Regression, Linear; Mean Difference (Final Values) = 0.09, 95% CI 2-sided [-0.13 to 0.31] — mean difference = (pain self-management) - (usual care)

14. Secondary Outcome: Prescription Opioid Misuse Index (POMI) Score
Description: as for outcome 13
Time Frame: 12 months after randomization
Population: as for outcome 13
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Pain Self-Management | Usual Care
Number analyzed (Participants) | 64 | 69
score on a scale | 0.39 [0.23 to 0.55] | 0.26 [0.11 to 0.41]
Statistical Analysis 1: Comparison: Pain Self-Management vs Usual Care; Test type: Equivalence — The null hypothesis is a point null of exactly 0 expected difference in POMI score between arms; p = 0.26, Regression, Linear; Mean Difference (Final Values) = 0.13, 95% CI 2-sided [-0.10 to 0.36] — mean difference = (pain self-management) - (usual care)

15. Secondary Outcome: Prescription Opioid Difficulties Scale (PODS) Score
Description: A 15-item questionnaire used to assess patient-perceived difficulties and concerns attributed to the use of opioid medication with scores between 0 and 60; higher scores indicate greater difficulties and concerns.
Time Frame: 6 months after randomization
Population: Randomized individuals with completed PODS questionnaires at 6- and/or 12-months post-randomization with non-missing baseline data used for adjustment in regression models.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Pain Self-Management | Usual Care
Number analyzed (Participants) | 61 | 67
score on a scale | 9.03 [1.71 to 16.36] | 7.43 [4.87 to 10.00]
Statistical Analysis 1: Comparison: Pain Self-Management vs Usual Care; Test type: Equivalence — The null hypothesis is a point null of exactly 0 expected difference in PODS score between arms; p = 0.54, Regression, Linear; Mean Difference (Final Values) = 1.60, 95% CI 2-sided [-3.47 to 6.66] — mean difference = (pain self-management) - (usual care)

16. Secondary Outcome: Prescription Opioid Difficulties Scale (PODS) Score
Description: as for outcome 15
Time Frame: 12 months after randomization
Population: as for outcome 15
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Pain Self-Management | Usual Care
Number analyzed (Participants) | 61 | 67
score on a scale | 8.15 [5.63 to 10.67] | 7.68 [5.08 to 10.27]
Statistical Analysis 1: Comparison: Pain Self-Management vs Usual Care; Test type: Equivalence — The null hypothesis is a point null of exactly 0 expected difference in PODS score between arms; p = 0.59, Regression, Linear; Mean Difference (Final Values) = 0.48, 95% CI 2-sided [-1.26 to 2.21] — mean difference = (pain self-management) - (usual care)

17. Secondary Outcome: Opioid Craving Score
Description: A single-item questionnaire used to assess opioid craving in the past week with scores between 0 and 10; higher scores indicate greater craving.
Time Frame: 6 months after randomization
Population: Randomized individuals with completed opioid craving questionnaires at 6- and/or 12-months post-randomization with non-missing baseline data used for adjustment in regression models.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Pain Self-Management | Usual Care
Number analyzed (Participants) | 64 | 71
score on a scale | 1.36 [0.79 to 1.93] | 1.40 [0.86 to 1.94]
Statistical Analysis 1: Comparison: Pain Self-Management vs Usual Care; Test type: Equivalence — The null hypothesis is a point null of exactly 0 expected difference in opioid craving score between arms; p = 0.90, Regression, Linear; Mean Difference (Final Values) = -0.04, 95% CI 2-sided [-0.66 to 0.57] — mean difference = (pain self-management) - (usual care)

18. Secondary Outcome: Opioid Craving Score
Description: as for outcome 17
Time Frame: 12 months after randomization
Population: as for outcome 17
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Pain Self-Management | Usual Care
Number analyzed (Participants) | 64 | 71
score on a scale | 0.97 [0.50 to 1.44] | 1.33 [0.74 to 1.91]
Statistical Analysis 1: Comparison: Pain Self-Management vs Usual Care; Test type: Equivalence — The null hypothesis is a point null of exactly 0 expected difference in PSEQ score between arms; p = 0.30, Regression, Linear; Mean Difference (Final Values) = -0.35, 95% CI 2-sided [-1.03 to 0.32] — mean difference = (pain self-management) - (usual care)

19. Secondary Outcome: At Least 30% Reduction in Daily Opioid Dose
Description: Indication of at least 30% reduction from baseline in the prior 30-day average prescribed morphine milligram equivalents (MME).
Time Frame: 6 months after randomization
Population: Randomized individuals with complete electronic pharmacy records during the 6- and/or 12-month post-randomization assessment period with non-missing baseline data used for adjustment in regression models.
Measure: Number; unit: participants
Arm/Group | Pain Self-Management | Usual Care
Number analyzed (Participants) | 72 | 76
participants | 9 | 4
Statistical Analysis 1: Comparison: Pain Self-Management vs Usual Care; Test type: Equivalence — The null hypothesis is a point null of the relative risk of 30% reduction from baseline equal exactly to 1; p = 0.20, Regression, Poison; Risk Ratio (RR) = 2.10, 95% CI 2-sided [0.68 to 6.53] — relative risk = (pain self-management)/(usual care)

20. Secondary Outcome: At Least 30% Reduction in Daily Opioid Dose
Description: as for outcome 19
Time Frame: 12 months after randomization
Population: as for outcome 19
Measure: Number; unit: participants
Arm/Group | Pain Self-Management | Usual Care
Number analyzed (Participants) | 72 | 76
participants | 10 | 7
Statistical Analysis 1: Comparison: Pain Self-Management vs Usual Care; Test type: Equivalence — The null hypothesis is a point null of the relative risk of 30% reduction from baseline equal exactly to 1; p = 0.53, Regression, Poison; Risk Ratio (RR) = 1.34, 95% CI 2-sided [0.54 to 3.32] — relative risk = (pain self-management)/(usual care)

ADVERSE EVENTS:
Time Frame: Data were collected for 12 months, ending at participants' final follow up time point.
Groups:
- Pain Self-Management: This arm includes patients Patients randomized to Pain self-management training; This intervention will have 4 components:
  1. telephone-delivered evidence-based pain self-management training,
  2. web-based video of successfully tapered patients with motivational interviewing debriefing,
  3. a voluntary, self-paced opioid taper
  4. opioid and non-opioid prescribing guidance for the patient's primary care provider.
Arm/Group | Pain Self-Management | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/79 | 0/74
Serious Adverse Events (participants affected / at risk) | 0/79 | 0/74
Other Adverse Events (participants affected / at risk) | 8/79 | 0/74
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pain Self-Management (N=79) | Usual Care (N=74)
Musculoskeletal pain after PMR (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0)
Headache after PMR (Nervous system disorders) | 2 (2) | 0 (0)
Stopped taking prescribed opioids (General disorders) | 1 (1) | 0 (0)
Increased anxiety / anger when reminded of appointment with study staff (Psychiatric disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-06-07): https://cdn.clinicaltrials.gov/large-docs/02/NCT03743402/Prot_SAP_000.pdf
  • Informed Consent Form (2020-05-14): https://cdn.clinicaltrials.gov/large-docs/02/NCT03743402/ICF_001.pdf